CLINICAL TRIAL: NCT04978389
Title: Inter-observer Reproductibility of Visual Estimation of Left Ventricular Ejection Fraction in Critical Care
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0462
Record Dates: First submitted 2021-07-19; First posted 2021-07-27 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Ventricular Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inter-observer reproductibility of visual estimation of left ventricular ejection fraction is known to be good in cardiology but has not been studied in ICU. The goal of the study is to determine if this reproductibility is good enough.

ELIGIBILITY:
Inclusion criteria:

* practitioners working in intensive care.
* age > 18 years

Exclusion criteria:

- Age under 18

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: practitioners working in intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
reproductibility of LVEF in percentage | day 1
  reproductibility of LVEF in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Kada KLOUCHE, MD PhD, Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC